CLINICAL TRIAL: NCT07151209
Title: A Prospective, Multicenter, Open-label Phase II Single-arm Clinical Trial Protocol on the Efficacy and Safety of Lparomlimab and Tuvonralimab in Combination With Lenvatinib and SOX Chemotherapy in Potentially Resectable MSI-H, dMMR Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma Patients
Brief Title: Immunotherapy Combined With Anti-angiogenic Therapy and Chemotherapy for Potentially Resectable MSI-H, dMMR Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-GasC-QIBA-3011
Record Dates: First submitted 2025-08-24; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma
Keywords: Iparomlimab and Tuvonralimab; lenvatinib; SOX
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab combination with lenvatinib and SOX (Experimental)
  Interventions: Drug: Iparomlimab and Tuvonralimab combined with lenvatinib and SOX

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab combined with lenvatinib and SOX — Iparomlimab and Tuvonralimab:5 mg/kg Q3W lenvatinib:8 mg/day orally SOX：oxaliplatin (130 mg/m² Q3W intravenous infusion), and S-1 (40 mg/m² BID orally on days 1-14)

SUMMARY:
Efficacy and safety of Iparomlimab and Tuvonralimab in combination with lenvatinib and SOX chemotherapy in potentially resectable MSI-H, dMMR locally advanced gastric or gastroesophageal junction adenocarcinoma patients: A prospective, multicenter, open-label Phase II single-arm clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and agree to comply with study requirements and the assessment schedule, and voluntarily sign the written informed consent form (ICF) before any trial-related procedures are implemented;
* Age greater than 18 years, regardless of gender. Histologically confirmed unresectable locally advanced or metastatic G/GEJ adenocarcinoma.
* No prior systemic treatment for unresectable locally advanced or metastatic G/GEJ adenocarcinoma. Previous neoadjuvant and/or adjuvant therapy is acceptable, but all systemic treatments must have been completed at least 6 months prior to the diagnosis of unresectable or metastatic disease.
* PD-L1 combined positive score (CPS) less than 1 as determined by tissue testing.
* At least one measurable lesion according to RECIST 1.1 criteria.
* ECOG performance status 0-1.
* Life expectancy >3 months.
* Adequate organ and marrow function:

Exclusion Criteria:

* 1. Known HER2-positive expression (immunohistochemistry [IHC] 3+ or 2+ with a fluorescence in situ hybridization HER2:CEP17 ratio ≥2).
* Presence of other malignancies within 5 years prior to treatment, with the exception of adequately treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, locally treated prostate cancer, and ductal carcinoma in situ (hormone therapy for non-metastatic prostate cancer or breast cancer is permitted).
* Known central nervous system metastases and/or carcinomatous meningitis.
* Patients with severe cardiac, pulmonary, hepatic, or renal dysfunction.
* Hypertension that cannot be controlled with antihypertensive medications (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg).
* History of bleeding within 4 weeks prior to screening, with any bleeding event graded as ≥3 according to CTCAE 5.0.
* Thrombotic events (arterial or venous) within 6 months prior to screening, such as cerebrovascular accident, deep vein thrombosis (excluding previously thrombosed veins deemed healed by the investigator), and pulmonary embolism.
* History of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation.
* Patients who have previously received anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies at any time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Up to approximately 2 years

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | Up to approximately 2 years
R0 resection rate | Up to approximately 2 years
Objective response rate (ORR) | Up to approximately 2 years
Event-free survival (EFS) | Up to approximately 2 years
12-month, 24-month, and 36-month event-free survival rates Disease-free survival (DFS) | Up to approximately 3 years
Overall survival (OS) | Up to approximately 5 years
12-month, 24-month, and 36-month overall survival rates | Up to approximately 3 years

IPD SHARING:
Plan to Share IPD: No